CLINICAL TRIAL: NCT04785924
Title: A Study Comparing Prospective Use of Imipenem/Cilastatin/Relebactam (IMI/REL) to Retrospective Data Using Meropenem/ Vabobactam (MVB) and Ceftazidime/Avibactam (CZA) in Treatment of Klebsiella Producing Carbapenemase Enterobacteriaceae Infections
Brief Title: Imipenem/Cilastatin/Relebactam (IMI/REL) in Treatment of CRE Infections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081742; MISP 59805 (Other: Atrium)
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2022-06

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection; KPC; Gram-Negative Bacterial Infections; Antibiotic Resistant Infection
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — imipenem, cilastatin and relebactam

STUDY DESIGN:
Intervention Model Description: A study of outcomes with use of an antibiotic, IMI/REL which can be compared with retrospective data of CRE-containing infections treated with MVB and CZA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Observation Treatment Group (Other): All patients observed while treated with IMI/REL.
  Interventions: Drug: Imipenem+Relebactam

INTERVENTIONS:
Drug: Imipenem+Relebactam — Antibiotic treatment for KPC producing CRE-containing gram-negative infections
  Other Names: Recarbrio

SUMMARY:
This is an observation study comparing prospective use of Imipenem/Cilastatin/Relebactam (IMI/REL) to retrospective data using Meropenem/Vabobactam (MVB)and Ceftazidime/Avibactam CZA) in treatment of Klebsiella Producing Carbapenemase Enterobacteriaceae infections at a tertiary care hospital. The objectives of the study are to demonstrate successful treatment of KPC containing Enterobacteriaceae infections with IMI/REL including in bacteremia, and to analyze treatment outcomes in use of IMI/REL for KPC-producing infections compared to historical clinical outcome data with CZA and MVB use at the same institution.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years of age) patients with a KPC-producing CRE infection at any site except for isolated urinary source. Patients may be initially enrolled once identified with a CRE infection defined as resistance to any carbapenem. Any carbapenem resistance will provide an initial mechanism of identifying study eligible patients in accordance with our institutions definition of CRE for infection prevention purposes. As this study is specific for KPC-producing CRE inclusion in the study analysis will require confirmation of a KPC gene by molecular analysis of the isolate and subjects enrolled may be subsequently removed from study and excluded from analysis if molecular testing reveals their CRE isolate to be a non-KPC mechanism of resistance. Polymicrobial infections at same or different sites can also be included as long as additional gram-negative active agents aside from IMI/REL are not needed for treatment.
2. Bacterial infection with Enterobacteriaceae excluding Morganellaceae
3. Ability and willingness to give informed consent. A Legal authorized representative may be used when the patient is unable to provide informed consent.
4. Be the first episode of a CRE infection to be treated with IMI/REL. Previously treatment with IMI/REL for a KPC-containing Enterobacteriaceae infection will exclude patients from enrollment.

Exclusion Criteria:

1. Receipt of more than 48 hours of effective antibiotic therapy against KPC containing infections (e.g. MVB, CZA) prior to first dose of IMI/REL being administered.
2. Infections localized to urinary source alone (bloodstream infections from urinary source will be included)
3. Infection with Morganellaceae
4. Prior serious allergic reaction to carbapenem therapy
5. Need for ongoing concomitant therapy with ganciclovir or valproic acid
6. Need for ongoing concomitant therapy with another antibiotic active against gram negative pathogens. Concomitant therapy with Vancomycin, Daptomycin, Linezolid, Clindamycin, Fidaxomicin, Nafcillin, Metronidazole, and Rifaximin will be allowed but no other antibiotic agents.
7. Pregnancy or ongoing breastfeeding. Women of childbearing age must test negative on a urine pregnancy test at time of screening for trial eligibility and remain either abstinent or use 2 forms of highly effective contraception for the duration of the IMI/REL administration during the study.
8. Inability to comply with study protocol or remain hospitalized for duration of study.
9. Life expectancy less than 72 hours in opinion of study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Clinical success | 30 days
  Clinical success defined as survival at 30 days, resolution of signs and symptoms of infection, sterilization of blood cultures within 7 days of treatment initiation in patients with bacteremia, and absence of recurrent infections.
Clinical success by site of infection | 30 days
  Clinical success in patients grouped by site of infection: bacteremia, respiratory, intra-abdominal infection, soft tissue, catheter associated and urinary tract. Subjects may be included in multiple groups if applicable for analysis.

SECONDARY OUTCOMES:
Mortality | 30 days
  Survival at 30 days
90 day Mortality | 90 days
  Survival at 90 days
Adverse effects | 90 days
  Incidence of nephrotoxicity, leukopenia, rash, hepatotoxicity, and seizure in treatment group
Total Length of hospital stays | 90 days
  Days of hospitalization for CRE infection
Recurrence of infection | 90 days
  Recurrence of CRE-containing infection within 90 days
Development of resistance | 90 days
  If recurrent CRE infection develops following index infection treated with IMI/REL, then incidence of IMI/REL resistance in subsequent bacterial cultures

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Polk, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-03-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04785924/ICF_000.pdf